CLINICAL TRIAL: NCT02764853
Title: Striving Towards EmPowerment and Medication Adherence (STEP-AD)
Acronym: STEP-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sannisha K Dale, Assistant Professor of Psychology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170281; 1K23MH108439 (NIH); 2016P001464 (Other: Mass General); 20170281 (Other: UMiami)
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: HIV
Keywords: HIV; Black; African American; Women; Cognitive Behavioral Therapy; Racism; Stigma; Discrimination; Gender related stressors; Resilience; Behavioral Medicine
MeSH Terms: conditions — Racism; Social Stigma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- STEP-AD (10 sessions) (Experimental): Participants in this arm will receive the manualized 10 session behavioral medicine intervention titled "Striving Towards EmPowerment and Medication Adherence".
  Interventions: Behavioral: Experimental Intervention (STEP-AD)
- Enhanced Treatment as Usual (E-TAU) (Active Comparator): Participants in this arm will receive 1 session of Lifesteps and appropriate services and referrals as needed, followed by bi-weekly check-ins with a study research assistant.
  Interventions: Behavioral: Enhanced Treatment as Usual (E-TAU)

INTERVENTIONS:
Behavioral: Experimental Intervention (STEP-AD) — This experimental intervention will consist of 10 sessions- 1 session of Lifesteps (problem solving for medication adherence) and 9 sessions of an intervention specifically tailored for Black women living with HIV to address trauma/abuse, racial discrimination, HIV stigma, and gender roles expectations in order to improve health outcomes (e.g., medication adherence, viral load), increase resiliency, and enhance adaptive coping strategies.
  Other Names: Striving Towards EmPowerment and Medication Adherence (STEP-AD)
  Arms: STEP-AD (10 sessions)
Behavioral: Enhanced Treatment as Usual (E-TAU) — Participants assigned to the E-TAU condition will receive 1 session of Lifesteps (problem solving for medication adherence) and appropriate services and referrals as needed
  Arms: Enhanced Treatment as Usual (E-TAU)

SUMMARY:
Striving Towards Empowerment and Medication Adherence (STEP-AD) is a research study aimed at developing an intervention for Black women living with HIV to address psychosocial factors (i.e. abuse/trauma histories, racial discrimination, HIV stigma/discrimination, and prescribed traditional gender roles) that have been associated with medication nonadherence or poor HIV outcomes (e.g. viral load, CD4), but are unaddressed in existing interventions.

DETAILED DESCRIPTION:
Among Black women with HIV in the U.S, generally low rates of adherence to ART are likely due to relevant psychosocial and contextual factors facing Black women with HIV, such as having a history of physical, sexual, and emotional abuse, post traumatic stress, racial discrimination, and contextual variables related to traditional gender roles; each of which are associated with worse HIV outcomes.

Despite the need, there is currently no evidenced-based psychosocial intervention for Black women with HIV that addresses these contextual factors to improve adherence to HIV self-care. A psychosocial intervention including content on reducing the effects of trauma and discrimination and increasing resilient coping strategies and gender empowerment may be most culturally appropriate, and therefore effective, in improving quality of life and increasing treatment adherence in Black women living with HIV/AIDS.

Striving Towards Empowerment and Medication Adherence (STEP-AD) is a research study aimed at developing an intervention for Black women living with HIV to address psychosocial factors (i.e. abuse/trauma histories, racial discrimination, HIV stigma/discrimination, and prescribed traditional gender roles) that have been associated with medication nonadherence or poor HIV outcomes (e.g. viral load, CD4), but are unaddressed in existing interventions.

Individual, in-depth qualitative interviews (n=30) were conducted with Black women with HIV and community stakeholders to gather information on the perceived acceptability and to inform the development of a manualized intervention of an integrated treatment to improve ART adherence by addressing trauma symptoms, racial discrimination, HIV discrimination, and gender related stressors experienced by Black women with HIV. This information was used to develop the resulting intervention.

An open pilot trial (n=5) of the resulting intervention was conducted (December 2015 through August 2016) in order to initially assess the feasibility of all study procedures and intervention delivery, acceptability, and a potential clinically significant improvement on ART adherence and hypothesized psychosocial mediators.

A pilot randomized control trial (RCT) comparing the newly developed intervention (N=25) to an enhanced treatment as usual control (N=25) on ART adherence (primary outcome) and viral load (secondary outcome) over 6 months (baseline, 10 weekly treatment visits [approximately 3 months], and a 6 month follow-up) begun enrolling participants as of August 2016.

Actual enrollment at baseline for all the phases are below. Please note that not all participants enrolled at baseline moved on to the relevant phase due the need to meet inclusion criteria.

Formative qualitative phase: 30 Black women living with HIV, 15 community Stakeholders

Open Pilot phase: 20 Black women living with HIV

Pilot RCT: 119 Black women living with HIV

Total: 184

ELIGIBILITY:
Inclusion Criteria:

1. HIV-positive
2. Identify as Black and/or African American
3. Age 18 or older
4. Biologically female
5. English speaking
6. Prescribed ART medication for at least the last two months
7. Low ART adherence (<80%) or detectable viral load within the past six months or
8. History of abuse/trauma (e.g. sexual, physical, and/or emotional abuse, experienced a traumatic event)
9. Capable of completing and fully understanding the informed consent process and the study procedures

Exclusion Criteria:

1. Significant mental health diagnosis requiring treatment (e.g., unstable bipolar disorder; any psychotic disorder)
2. Inability (e.g., due to cognitive or psychiatric difficulties) or unwillingness to provide informed consent
3. Recent (past 6 months) behavioral treatment for ART adherence or trauma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-12; Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
ART Medication Adherence | Change from Baseline until study completion (~ 9 months)
  Adherence to antiretroviral therapy (ART) as captured by the Wisepill electronic adherence monitor. Change from baseline adherence.

SECONDARY OUTCOMES:
HIV Viral Load | Change from Baseline until study completion (~ 9 months)
  A decrease in participants' HIV viral load ( and/or a change from detectable to undetectable) since the study's start as captured via medical records or blood specimen if recent medical records are unavailable.
Trauma Symptoms | Change from Baseline until study completion (~ 9 months)
  A decrease in participants' trauma symptoms since the study's start as captured by the Davidson Trauma Scale (DTS), a 17-item self-rating scale used to assess symptoms of Post-Traumatic Stress Disorder (PTSD).

CONTACTS AND LOCATIONS:
Overall Officials: Sannisha K Dale, PhD, EdM, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dale SK, Pierre-Louis C, Bogart LM, O'Cleirigh C, Safren SA. Still I rise: The need for self-validation and self-care in the midst of adversities faced by Black women with HIV. Cultur Divers Ethnic Minor Psychol. 2018 Jan;24(1):15-25. doi: 10.1037/cdp0000165. Epub 2017 Jun 12. PMID 28604021
- [Result] Dale SK, Safren SA. Striving Towards Empowerment and Medication Adherence (STEP-AD): A Tailored Cognitive Behavioral Treatment Approach for Black Women Living With HIV. Cogn Behav Pract. 2018 Aug;25(3):361-376. doi: 10.1016/j.cbpra.2017.10.004. Epub 2017 Dec 5. PMID 30147289
- [Derived] Boga DJ, Juste RS, Etienne K, Dale SK. Using network analysis to elucidate the relationships among support systems, trauma and depressive symptoms, self-silencing, and risk of HIV viral non-suppression among black women living with HIV. J Behav Med. 2025 Apr;48(2):268-279. doi: 10.1007/s10865-024-00530-1. Epub 2024 Nov 23. PMID 39580576
- [Derived] Reid R, Dale SK. Structural equation modeling of microaggressions, religious and racism-related coping, medication adherence, and viral load among Black women living with HIV. J Behav Med. 2023 Oct;46(5):837-848. doi: 10.1007/s10865-023-00403-z. Epub 2023 Mar 30. PMID 36997766
- [Derived] Boga DJ, Dale SK. Black Women Living with HIV: A Latent Profile Analysis of Intersectional Adversities, Resilience, and Mental Health. AIDS Patient Care STDS. 2022 Sep;36(9):364-374. doi: 10.1089/apc.2022.0053. Epub 2022 Aug 30. PMID 36040393